CLINICAL TRIAL: NCT06818305
Title: A Multicenter, Open-Label, Factorial Design, Randomized Controlled Study to Explore the Efficacy and Safety of Finerenone and Empagliflozin, Alone or in Combination, in Delaying Renal Function Progression in High-Risk CKD Patients After Radical Nephrectomy for Renal Cell Carcinoma
Brief Title: Efficacy and Safety of Finerenone and Empagliflozin in Delaying Renal Function Progression After Radical Nephrectomy in High-Risk CKD Patients: A Multicenter RCT
Acronym: EmFin-Nx
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The patient enrollment rate is proceeding too slowly
Sponsor: Jinling Hospital, China (Other)
Collaborators: The Affiliated Hospital of Xuzhou Medical University (Other); Qilu Hospital of Shandong University (Other); Yantai Yuhuangding Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Le Qu, Associate chief urologist, Jinling Hospital, China
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2024DZKY-097-02
Record Dates: First submitted 2025-01-28; First posted 2025-02-10 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-02

CONDITIONS: Renal Cell Carcinoma (Kidney Cancer); Renal Cell Carcinoma (RCC); Nephrectomy; Chronic Kidney Disease(CKD)
Keywords: Renal Cell Carcinoma; Radical Nephrectomy; Chronic Kidney Disease; Renal Functional Compensation; Finerenone; Empagliflozin; Renal Protection; Clinically Significant CKD; Randomized Controlled Trial; Mineralocorticoid Receptor Antagonist; CKD; RCC; MRA; csCKD; RCT
MeSH Terms: conditions — Carcinoma, Renal Cell; Kidney Neoplasms; Renal Insufficiency, Chronic | interventions — finerenone; empagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Finerenone (Experimental): Participants will receive finerenone.
  Interventions: Drug: Finerenone (BAY 94-8862)
- Empagliflozin (Experimental): Participants will receive empagliflozin.
  Interventions: Drug: Empagliflozin 10 mg
- Combination therapy of Finerenone and Empagliflozin (Experimental): Participants will receive finerenone and empagliflozin.
  Interventions: Drug: Finerenone (BAY 94-8862); Drug: Empagliflozin 10 mg
- Blank control group (No Intervention): Participants did not receive medication.

INTERVENTIONS:
Drug: Finerenone (BAY 94-8862) — Adjusting lifestyle and managing underlying conditions according to the "Chronic Kidney Disease Early Screening, Diagnosis, and Prevention Guidelines (2022 Edition)" + Finerenone (10mg/d or 20mg/d).
  Arms: Combination therapy of Finerenone and Empagliflozin; Finerenone
Drug: Empagliflozin 10 mg — Adjusting lifestyle and managing underlying conditions according to the "Chronic Kidney Disease Early Screening, Diagnosis, and Prevention Guidelines (2022 Edition)" + Empagliflozin (10mg/d).
  Arms: Combination therapy of Finerenone and Empagliflozin; Empagliflozin

SUMMARY:
The goal of this clinical trial is to evaluate whether Finerenone and Empagliflozin, either alone or in combination, can delay the progression of renal function decline in patients at high risk for chronic kidney disease (CKD) following radical nephrectomy for renal cell carcinoma (RCC). It will also assess the safety of these treatments.The main questions it aims to answer are:

1. Does Finerenone and Empagliflozin, alone or in combination, slow the progression of renal function decline in high-risk CKD patients after RCC surgery?
2. What are the safety profiles of Finerenone and Empagliflozin in this patient population?

Researchers will compare the treatment groups (Finerenone and Empagliflozin) to a blank control group (no drug) to determine if the treatments effectively delay renal function decline.

Participants will:

1. Take either Finerenone and Empagliflozin (alone or in combination) or a blank control every day for 1 years.
2. Visit the clinic once every 3 months for checkups and tests.
3. Track their eGFR and other kidney function markers regularly.
4. Keep a diary to record any adverse events or changes in their health condition during the study.

DETAILED DESCRIPTION:
The "three-high" state (high pressure, high perfusion, and high filtration) within the glomerulus is a major contributor to the progression of chronic kidney disease (CKD). After nephrectomy for renal cell carcinoma (RCC), patients experience significant loss of nephrons in the affected kidney within a short period. In response, the remaining nephrons begin compensatory work under high load conditions, leading to increased glomerular filtration rate (GFR, high filtration), elevated plasma flow (high perfusion), and increased capillary transmembrane pressure (high pressure). This places patients at a higher risk for acute kidney injury (AKI) and CKD. The afferent and efferent arterioles are two critical vessels in the glomerulus, playing a pivotal role in the kidney's filtration process. The afferent arteriole delivers blood into the glomerulus, while the efferent arteriole carries blood out, entering the renal tubular system. During the compensatory phase following nephron loss, the afferent arteriole of the residual nephrons dilates more significantly than the efferent arteriole, leading to increased blood flow into the glomerulus and thus contributing to the "three-high" state of the kidney.

The "three-high" state was traditionally considered an adaptive change in the kidney under both physiological and pathological conditions, involving changes in renal hemodynamics, glomerular hypertrophy, afferent arteriole dilation, and efferent arteriole constriction. Under these conditions, glomerular enlargement occurs, which in turn stretches mesangial cells, leading to the excessive production and accumulation of extracellular matrix (ECM). This exacerbates glomerular damage, eventually progressing to irreversible glomerulosclerosis.

The salt intake in the Chinese population is significantly higher than the levels recommended by the World Health Organization (WHO). High salt intake significantly elevates the risk of CKD, representing the most prominent external factor contributing to glomerular hypertension. Thus, high-salt diets are a major risk factor for the progression of chronic kidney disease. High salt intake induces increased local renin-angiotensin-aldosterone system (RAAS) activity in the kidneys, promoting inflammation, fibrosis, and oxidative stress, all of which contribute to kidney damage. Moreover, overactivation of the mineralocorticoid receptor (MR) exacerbates glomerular efferent arteriole constriction, leading to higher glomerular capillary pressure, glomerular capillary sclerosis, and reduced vascular compliance. These conditions further aggravate the "three-high" state of the kidney in patients who have undergone nephrectomy, increasing the risk of post-surgical CKD. Furthermore, the Asian population is more likely to have genetic predispositions for salt sensitivity, and both salt sensitivity and high salt intake can lead to excessive MR activation, increasing the risk of CKD.

After radical nephrectomy, patients with renal cell carcinoma are at significantly increased risk for CKD, yet accurate prediction of long-term CKD development remains challenging. Although many studies have assessed post-operative renal function changes, validated clinical tools are limited, with most unable to accurately predict renal function outcomes after nephrectomy. Additionally, international guidelines offer limited recommendations on the post-operative CKD risk, with follow-up plans primarily focused on cancer recurrence risk and less on renal function changes.

Renal functional compensation (RFC) and split renal function (SRF) are crucial for maintaining overall renal function after radical nephrectomy for RCC. RFC refers to the ability of the remaining kidney tissue to increase its filtration rate to compensate for the loss of renal function. RFC typically begins within two weeks post-surgery, with compensation reaching up to 10%, peaking at around three months post-surgery (compensation rate of 26%), and stabilizing by the fifth year post-surgery. SRF plays an important role in predicting renal function after nephrectomy; it is measured through pre-operative imaging to assess the proportion of renal function between the two kidneys. Pre-operative SRF and GFR values can help predict the post-operative new baseline GFR (NB-GFR). A prediction formula based on SRF and pre-operative GFR has been validated and is highly accurate for estimating post-operative NB-GFR.This formula has been proven to provide accurate predictions for post-surgical renal function recovery. Additionally, Robert J et al. developed and validated a clinically significant CKD (csCKD) scoring system, based on routine clinical variables, to stratify the risk of significant CKD occurrence within 12 months after nephrectomy. This scoring system is simple and reliable, aiding clinicians in early identification and intervention for high-risk patients, optimizing post-operative management. We have conducted a multicenter clinical study to validate the predictive capability of the csCKD score, but for high-risk patients identified by this score, there remains a lack of effective intervention strategies to prevent or reduce the long-term development of CKD. Therefore, further studies are needed to explore potential interventions.

Finerenone is a non-steroidal, selective mineralocorticoid receptor antagonist (MRA). MR is widely expressed in various tissues, including podocytes, macrophages, mesangial cells, fibroblasts, and epithelial cells in the kidneys, as well as in cardiac myocytes, macrophages, fibroblasts, endothelial cells, and vascular smooth muscle cells in the cardiovascular system. When MR is overactivated, it induces a series of pathophysiological changes in the kidney and heart, including inflammation, fibrosis, myocardial hypertrophy, apoptosis, sodium and water retention, and vasoconstriction. MR activation is influenced by multiple factors, including increased ACTH, endothelin-1, elevated K+, decreased Na+, and RAAS activation, which induce aldosterone secretion, thereby enhancing MR activation. In certain circumstances, glucocorticoid elevation can also activate MR. Traditional RAAS inhibitors (RASi) block only the MR activation induced by RAAS, but they fail to comprehensively inhibit MR overactivation, with 40-53% of patients developing aldosterone escape, leading to increased serum aldosterone levels despite RASi therapy. Finerenone, as a selective MRA, directly antagonizes MR, achieving comprehensive inhibition of MR overactivation. In the kidneys, Finerenone dilates the efferent arteriole of the glomerulus, reducing glomerular blood flow, thus alleviating the "three-high" state and slowing renal aging or damage. Additionally, Finerenone binds to MR in a way that prevents conformational changes and the recruitment of transcriptional co-regulatory factors, blocking the inflammatory and fibrotic gene expression induced by MR overactivation, reducing kidney and heart inflammation and fibrosis.

Finerenone has a stronger ability than traditional steroidal MRAs to block MR co-activation and induce co-repressor factor binding, thus effectively suppressing renal inflammation and fibrosis. Unlike steroidal MRAs, Finerenone significantly reduces the occurrence of sex hormone-related adverse effects and hyperkalemia, making it a safer alternative.

Empagliflozin is a selective sodium-glucose cotransporter-2 (SGLT-2) inhibitor, primarily acting on the S1 segment of the proximal convoluted tubule in the kidney. SGLT-2 is a high-capacity, low-affinity transporter responsible for the reabsorption of glucose and sodium ions from the urine into the bloodstream. Empagliflozin inhibits SGLT-2, significantly reducing the reabsorption of glucose and sodium, which lowers blood glucose levels and promotes osmotic diuresis and sodium excretion. This process reduces blood volume and cardiac load, providing dual benefits for the cardiovascular and renal systems. The renal protective effects of SGLT-2 inhibitors are multifaceted, including improving glomerular hyperfiltration, reducing proteinuria, alleviating renal hypoxia, lowering uric acid levels, and mitigating inflammation and oxidative stress. In patients undergoing radical nephrectomy, increased glomerular blood flow can be mitigated by SGLT-2 inhibitors, which reduce sodium and glucose reabsorption, raising sodium concentration in the macula densa and activating tubuloglomerular feedback to constrict the afferent arteriole, thus mitigating the hyperfiltration state. Additionally, SGLT-2 inhibitors such as Empagliflozin protect the kidneys by reducing inflammation and oxidative stress.

The FIDELIO-DKD study demonstrated that Finerenone reduces the risk of renal composite outcomes by 18% and cardiovascular composite outcomes by 14% in patients with diabetes and CKD. After four months of treatment, Finerenone reduced urinary albumin-to-creatinine ratio (UACR) by 31%. The FIGARO-DKD study confirmed that Finerenone reduces the risk of cardiovascular composite outcomes by 13% in diabetes-associated CKD patients. Asian patients showed greater renal and cardiovascular benefits with Finerenone compared to the overall population. According to the FIDELIO-DKD study, Finerenone reduced the risk of renal composite outcomes by 41% and cardiovascular composite outcomes by 25% in Chinese patients, showing superior renal and cardiovascular benefits compared to the global population. Consequently, Finerenone became the first MRA to be approved globally for the treatment of type 2 diabetes-related kidney disease, with approval in the U.S. (July 2021), the EU (February 2022), Japan (February 2022), and China (June 2022). It is indicated for the treatment of adult chronic kidney disease patients with type 2 diabetes, reducing the risk of progressive decline in eGFR and end-stage renal disease, thus providing renal protection.

Regarding SGLT2 inhibitors, several large-scale clinical trials (e.g., DAPA-CKD, EMPA-KIDNEY, CANVAS, DECLARE-TIMI58) have demonstrated that SGLT-2 inhibitors not only effectively lower blood glucose but also provide significant renal protection. In the EMPA-KIDNEY phase III trial, Empagliflozin significantly reduced the incidence of renal and cardiovascular adverse events in CKD patients. Compared to placebo, Empagliflozin reduced the risk of the primary composite endpoint (eGFR decline ≥50%, end-stage renal disease, or death from renal or cardiovascular causes) by 39%. In terms of renal function protection, the Empagliflozin group had an annual mean eGFR decline rate of -2.86 mL/min/1.73m², whereas the placebo group had -3.79 mL/min/1.73m², demonstrating significant slowing of progression. Empagliflozin showed efficacy and safety in CKD patients, regardless of type 2 diabetes status. Furthermore, recent reports have shown that the renal and cardiovascular protective effects of Empagliflozin persist for up to 12 months after discontinuation in patients with progressive CKD.

Currently, several clinical studies are ongoing regarding Finerenone and Empagliflozin in different patient populations. The FIND-CKD study is evaluating the efficacy and safety of adding Finerenone to standard therapy for non-diabetic CKD, with a target completion date of November 2025. The EFFEKTOR study aims to assess the feasibility, tolerance, efficacy, and safety of Finerenone in kidney transplant recipients (KTR), with a target completion date of December 2025. The Empagliflozin in ESKD study explores the use of Empagliflozin in end-stage kidney disease patients to expand its indications and evaluate its efficacy in different populations. A real-world study in China involving 58 patients undergoing radical nephrectomy and receiving Finerenone treatment found no patients discontinuing the drug due to adverse events, with efficacy still under follow-up evaluation.

Based on the mechanisms of kidney injury following RCC surgery, coupled with the selective blockade of MR by Finerenone and SGLT-2 inhibition by Empagliflozin, which alleviate the "three-high" state of the kidney and exert anti-inflammatory and anti-fibrotic effects, we plan to conduct a multicenter, open-label, randomized controlled trial to evaluate the efficacy and safety of Finerenone and Empagliflozin, alone or in combination, in delaying the progression of renal dysfunction in high-risk (csCKD ≥7) patients with localized kidney tumors (T1-T2) following radical nephrectomy. This study aims to provide timely renal protection strategies for high-risk patients susceptible to post-surgical CKD.

ELIGIBILITY:
Inclusion Criteria:

* 1、Voluntary participation in the study and signing of the informed consent form, with the ability to comply with the study or follow-up procedures.

  2、Age ≥ 18 years (at the time of signing the informed consent form), regardless of sex.

  3、Patients with renal tumors (T1-T2) who are scheduled to undergo radical nephrectomy; no specific surgical procedure requirements.

  4、Normal imaging of the healthy kidney at screening. 5、csCKD score ≥ 7 (moderate risk: 7-8 points; high risk: 9-10 points). 6、Preoperative difference in renal function of <10% (healthy kidney function - affected kidney function).

  7、Serum potassium ≤ 5.0 mmol/L. 8、Urinary albumin-to-creatinine ratio (UACR) < 30 mg/g (3 mg/mmol). 9、ECOG performance status score of 0-2. 10、Normal cardiovascular, pulmonary, and liver function. 11、Women of non-reproductive potential are not required to undergo pregnancy testing or provide consent for appropriate contraceptive use. Non-reproductive potential is defined as women who have undergone hysterectomy, bilateral salpingectomy, oophorectomy, or are postmenopausal (with no other medical reasons for amenorrhea for 12 months).

  12、Women of reproductive potential must have a negative urine or serum pregnancy test within 7 days prior to enrollment, and must agree to use appropriate contraception during the study and for 8 weeks after the last dose of study intervention. Appropriate contraception is defined as an intrauterine device (IUD) or physical barriers (e.g., condoms)

Exclusion Criteria:

* Patients who meet any of the following conditions:

  1. Preoperative eGFR < 60 mL/min/1.73m² (calculated using the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation).
  2. eGFR of the healthy kidney < 30 mL/min/1.73m².
  3. Type 1 diabetes (T1D) or diabetic ketoacidosis.
  4. Pregnant or breastfeeding women.
  5. Patients with a desire to conceive during the study period or within 2 months after the study; male patients planning to conceive or donate sperm during the study period or within 3 months after the study.
  6. Body mass index (BMI) < 18.5 kg/m² or > 30 kg/m².
  7. Previous or concurrent participation in another clinical study (≤30 days before randomization).
  8. Communication disorders preventing full understanding or cooperation, or poor compliance.
* Patients with the following medical or surgical history:

  1. Urological structural abnormalities or unresolved functional abnormalities (e.g., duplicated kidney, polycystic kidney, horseshoe kidney, solitary kidney, renal artery stenosis, urinary tract obstruction, kidney stones, benign prostatic hyperplasia, prostatitis, or previous kidney surgery, etc.), long-term catheterization, etc.
  2. History of or planned kidney replacement therapy (dialysis or kidney transplant) within 12 weeks or kidney transplant planned within 12 months.
  3. Uncontrolled blood glucose: HbA1c ≥ 12%.
  4. Uncontrolled blood pressure: Initial or follow-up seated systolic blood pressure (SBP) ≥ 180 mmHg or seated diastolic blood pressure (DBP) ≥ 110 mmHg, or symptomatic hypotension and/or systolic blood pressure < 90 mmHg, or clinically judged hypovolemic patients.
  5. Previous radiation therapy or ablation therapy to the healthy kidney or other surgical procedures.
  6. History of heart failure (NYHA Class III-IV) or hospitalization due to fluid retention.
  7. Clinical history of cerebrovascular disease (transient ischemic attack or stroke) or coronary artery disease (hospitalization for myocardial infarction or unstable angina, new-onset angina, or coronary angiography showing stenosis, coronary artery revascularization) within the last 6 months.
  8. History of pulmonary hypertension, pulmonary fibrosis, or any lung condition requiring oxygen therapy (e.g., chronic obstructive pulmonary disease, emphysema).
  9. Severe peripheral edema or facial edema within 4 weeks of screening, requiring diuretic treatment, or history of myxedema.
  10. Liver function impairment, with any of the following: history of hepatic encephalopathy, esophageal varices, portal vein shunt surgery, severe liver dysfunction (Child-Pugh Class C), ALT or AST > 3 times the upper limit of normal (ULN), or total bilirubin > 2 times the ULN at screening.
  11. Primary adrenal insufficiency (Addison's disease).
  12. Recurrent urinary tract infections within the past 6 months.
  13. Organ or bone marrow transplant history.
  14. History of malignancy, except for those with: cured or in remission for ≥5 years, or radically excised basal cell carcinoma, squamous cell carcinoma, or any in situ carcinoma at any site.
  15. Received cytotoxic drugs, immunosuppressive therapy, or other immunotherapy for primary or secondary kidney disease within the last 6 months.
  16. Hematocrit ≤ 30%.
  17. Conditions that may significantly affect drug absorption, distribution, metabolism, or excretion, including but not limited to: 1) active inflammatory bowel disease in the last 6 months; 2) history of gastric surgery (e.g., gastrectomy, gastrointestinal anastomosis, or bowel resection); 3) history of gastrointestinal ulcers and/or gastrointestinal or rectal bleeding in the last 6 months; 4) history of pancreatic injury or pancreatitis in the last 6 months.
  18. Other complex medical conditions that may interfere with the study behavior or increase risks, such as organ failure, immunodeficiency diseases or HIV-positive status, viral hepatitis, cognitive disorders, or severe physical or mental illnesses.
  19. Any disease with a life expectancy of less than 12 months.
  20. Known allergy to the study drug or any drugs with a similar chemical structure or excipients. Note: Finerenone contains lactose; patients with galactose intolerance or malabsorption, or lactase deficiency are contraindicated.
* Current or past use of the following medications:

  1. Currently using potassium-sparing diuretics (e.g., amiloride, triamterene), other mineralocorticoid receptor antagonists (e.g., eplerenone, esaxerenone, spironolactone, canrenone), and unable to stop the medication ≥ 4 weeks before screening.
  2. Strong CYP3A4 inhibitors or inducers (e.g., itraconazole, ketoconazole, ritonavir, nelfinavir, cobicistat, telithromycin, naftifine, or grapefruit/grapefruit juice), and unable to stop at least 7 days before randomization.
  3. Currently receiving systemic treatment for malignancy.
  4. History of drug or alcohol abuse within the last 12 months.
  5. Received Empagliflozin treatment within 8 weeks prior to dosing or known intolerance to Empagliflozin.
  6. Received Finerenone treatment within 12 months prior to dosing.
  7. Kidney transplant patients or those on high-dose steroids or immunosuppressive therapy (e.g., systemic lupus erythematosus, ANCA-associated vasculitis, glomerulonephritis, nephrotic syndrome).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
The incidence of CKD stage 3b (eGFR < 45 mL/min/1.73m²) at 1 year post-surgery | 1 year after surgery

SECONDARY OUTCOMES:
The safety and tolerability of Finerenone and Empagliflozin, alone or in combination | Up to end of study visit (up to approximately 12 months)
  The incidence of hyperkalemia、hypotension、Urinary system infection and hypoglycemia
Renal function compensation rate 1 year after surgery | 1 year after surgery
The change rate in the volume of the healthy kidney parenchyma at 1 year post-surgery | 1 year after surgery
Rate of change of normal unit renal parenchymal function at 1 year after surgery | 1 year after surgery
The incidence of UACR ≥ 30 mg/g at 1 year post-surgery. | 1 year after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Jinling Hospital, Affiliated Hospital of Medical School, Nanjing University, Nanjing, Nanjing, Jiangsu, China